CLINICAL TRIAL: NCT02545179
Title: Ethics Committee of the University of Social Welfare and Rehabilitation Science
Brief Title: Web-based Daily Care Training of Children With Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Social Welfare and Rehabilitation Science (Other)
Responsible Party: Principal Investigator, Zahra Nobakht, PhD student, occupational therapy department,University of Social Welfare and Rehabilitation Science, University of Social Welfare and Rehabilitation Science
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IR.USWR.REC.1394.111
Record Dates: First submitted 2015-09-07; First posted 2015-09-09 (Estimated); Last update posted 2015-09-10 (Estimated); Status verified 2015-09

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intervention (Experimental): web-based daily care training 12 week interactive web based caring training education
  Interventions: Other: web-based daily care training
- control (No Intervention): Previous therapy

INTERVENTIONS:
Other: web-based daily care training — 12 week interactive web based caring training education
  Arms: intervention

SUMMARY:
Purpose:Effect of web-based daily care training on the quality of life of caregivers of children with cerebral palsy.

study design: Single-blind clinical trial. study population: Caregivers of children with cerebral palsy. Inclusion criteria: caregiver -Mother of a child with cerebral palsy who spent most time on child care- Children with cerebral palsy aged 4 to 12 years old living in Alborz province that clinical diagnosis of cerebral palsy registered in their clinical records. Moderate and severe cerebral palsy (gross motor function levels 3 to 5). caregiver have facilities and basic knowledge of using Internet (Declared access to the Internet at least one hour a week). exclusion criteria: taking care of two or more children with disability. participated in previous face to face training programs.

Sample size: 100. Intervention: Web-based daily care training. intervention time: 12-week. Outcome of the study: the quality of life of caregivers

DETAILED DESCRIPTION:
step1: web development and design

1. development of educational content (4 weeks)
2. Create a paper version of the site (2 weeks)
3. Create a web-based version of the site (4 weeks)
4. pilot study (6 weeks) step 2: RCT (12 weeks)

ELIGIBILITY:
Inclusion Criteria:

* caregiver_ Mother of a child with cerebral palsy who spent most time on child care Children with cerebral palsy aged 4 to 12 years old living in Alborz province that clinical diagnosis of cerebral palsy registered in their clinical records
* Moderate and severe cerebral palsy (gross motor function levels 3 to 5)
* caregiver have facilities and basic knowledge of using Internet (Declared access to the Internet at least one hour a week)

Exclusion Criteria:

* taking care of two or more children with disability
* participated in previous training programs

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-01 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
quality of life of caregivers | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Zahra Nobakht, PhD student, Principal Investigator — Occupational therapy department, University of Social Welfare and Rehabilitation Sciences